CLINICAL TRIAL: NCT06052956
Title: A Phase 2 Study to Assess Efficacy of Methylene Blue Photodynamic Therapy for Treatment of Deep Tissue Abscesses
Brief Title: Efficacy of Methylene Blue Photodynamic Therapy for Treatment of Deep Tissue Abscesses
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Timothy Baran, Assistant Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00008702
Record Dates: First submitted 2023-09-18; First posted 2023-09-25 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Abscess
Keywords: Abscess; Drainage; Photodynamic Therapy
MeSH Terms: conditions — Abscess | interventions — Methylene Blue; Fat Emulsions, Intravenous

STUDY DESIGN:
Intervention Model Description: The study includes three arms: (1) MB-PDT at a fixed drug/light dose plus standard of care abscess drainage, (2) MB-PDT at a patient-specific dose determined by pre-treatment optical measurements plus standard of care abscess drainage, and (3) standard of care abscess drainage.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The subject and study doctor will not be masked to group assignment, as it would be difficult or impossible to do so and unethical to subject patients to sham procedures if they are not assigned to a PDT group. However, all follow-up and subsequent data collection will be performed by a member of the study team that is masked to group assignment. Group assignment will only be unmasked to the study biostatistician at the time of statistical analysis. The remainder of the study team will only be unmasked after final results are published. This will reduce the potential for bias in collection of follow-up data, and protect the integrity of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- MB-PDT at pre-defined dose plus standard of care abscess drainage (Experimental): Each subject in this arm will receive standard of care abscess drainage, methylene blue, lipid emulsion, and laser illumination at an optical power defined by their abscess size.
  Interventions: Drug: Methylene Blue; Drug: Lipid Emulsion; Device: Insertion of optical fiber; Device: Laser Illumination (pre-defined dose); Procedure: Standard of care abscess drainage
- MB-PDT at patient-specific dose plus standard of care abscess drainage (Experimental): Each subject in this arm will receive standard of care abscess drainage, methylene blue, lipid emulsion, optical spectroscopy, and laser illumination. The optical power for laser illumination will be determined by their abscess morphology and the results of optical spectroscopy.
  Interventions: Drug: Methylene Blue; Drug: Lipid Emulsion; Device: Insertion of optical fiber; Device: Optical Spectroscopy Measurement; Device: Laser Illumination (patient-specific dose); Procedure: Standard of care abscess drainage
- Standard of care abscess drainage (Other): Each subject in this arm will receive standard of care abscess drainage
  Interventions: Procedure: Standard of care abscess drainage

INTERVENTIONS:
Drug: Methylene Blue — Administration of 0.1 mg/mL methylene blue to the abscess cavity, followed by a 10 minute incubation interval. After this incubation interval, the methylene blue solution will be aspirated from the cavity and flushed twice with sterile saline.
  Other Names: Methylene Blue Injection, 1%
  Arms: MB-PDT at patient-specific dose plus standard of care abscess drainage; MB-PDT at pre-defined dose plus standard of care abscess drainage
Drug: Lipid Emulsion — The abscess cavity will be filled with sterile 0.1% lipid emulsion solution to gently distend the cavity and, through efficient light scattering, to homogenize the light dose to the walls of the cavity. After laser illumination, the Intralipid will be aspirated from the cavity.
  Other Names: Intralipid 20%; Nutrilipid 20%
  Arms: MB-PDT at patient-specific dose plus standard of care abscess drainage; MB-PDT at pre-defined dose plus standard of care abscess drainage
Device: Insertion of optical fiber — A sterile, FDA-approved optical fiber will be advanced to the approximate center of the abscess cavity via the drainage catheter under image guidance. Following laser illumination, the fiber will be withdrawn.
  Other Names: Boston Scientific Flexiva Pulse ID
  Arms: MB-PDT at patient-specific dose plus standard of care abscess drainage; MB-PDT at pre-defined dose plus standard of care abscess drainage
Device: Laser Illumination (pre-defined dose) — Laser illumination will be delivered via the optical fiber for a duration of 20 minutes. The optical power will be set such that the fluence rate at the abscess wall due to ballistic photons is 20 mW/cm2.
  Other Names: Modulight ML7710 Laser System
  Arms: MB-PDT at pre-defined dose plus standard of care abscess drainage
Device: Optical Spectroscopy Measurement — The same sterile optical fiber used for treatment will be advanced through the drainage catheter/needle in order to make gentle contact with the wall of the cavity. Low-intensity, polarized white light will be delivered by a tungsten halogen lamp by the fiber, and captured by the same fiber. Light that has been de-polarized by interaction with tissue will be detected by a spectrometer and analyzed to extract tissue optical properties. Upon completion of these measurements, the fiber optic will be withdrawn, gently wiped with sterile gauze, and returned to the procedure cart.
  Arms: MB-PDT at patient-specific dose plus standard of care abscess drainage
Device: Laser Illumination (patient-specific dose) — Laser illumination will be delivered via the optical fiber for a duration of 20 minutes. The optical power will be set to deliver a fluence rate of 20 mW/cm2 in 95% of the abscess wall, based upon abscess morphology and optical spectroscopy results.
  Other Names: Modulight ML7710 Laser System
  Arms: MB-PDT at patient-specific dose plus standard of care abscess drainage
Procedure: Standard of care abscess drainage — Following standard practice, a drainage catheter will be placed in the abscess cavity and used to aspirate purulent fluid.
  Other Names: Image-guided percutaneous drainage

SUMMARY:
The objective of this Phase 2 study is to evaluate the efficacy of methylene blue photodynamic therapy (MB-PDT) performed at the time of percutaneous abscess drainage for disinfection of deep tissue abscesses. The study includes three arms: (1) MB-PDT at a fixed drug/light dose plus standard of care abscess drainage , (2) MB-PDT at a patient-specific dose determined by pre-treatment optical measurements plus standard of care abscess drainage , and (3) standard of care abscess drainage. The primary endpoint is reduction in time to removal of the drainage catheter.

DETAILED DESCRIPTION:
Abscesses form as a result of the interaction between an acute microbial infection and the host immune system, and generally result in fever, nausea, and acute abdominal pain. If untreated, the mortality rate can be high. Abscesses are routinely managed by image-guided percutaneous drainage and delivery of systemic antibiotics. Despite this standard of care, abscesses remain a significant source of morbidity, mortality, and hospital stay. Further, response can vary widely between patients. Many abscesses also contain antibiotic resistant species.

Photodynamic therapy (PDT), which relies upon the combination of photosensitive dyes known as photosensitizers, excitation by visible light, and molecular oxygen to generate cytotoxic reactive oxygen species, represents a powerful adjunct to standard of care drainage. A Phase 1 clinical trial aimed at assessing the safety and feasibility of methylene blue (MB) PDT at the time of percutaneous abscess drainage (ClinicalTrials.gov Identifier: NCT02240498) was completed. No adverse or serious adverse events were observed, and the procedure was well tolerated by all subjects. Based on these encouraging Phase 1 results, the current study therefore aims to assess efficacy of MB-PDT by quantification of time to removal of the drainage catheter and microbiological analysis of pre- and post-PDT aspirate samples.

This is a single center, randomized, open-label Phase 2 clinical trial, which will be conducted in accordance with the principles of good clinical practice and following approval by both the FDA and local IRB. Patients who have been diagnosed with a drainable abscess, that meet all inclusion/exclusion criteria, and have the approval of their primary care team, will be offered enrollment in the study. Consented subjects will be assigned prospectively to one of three arms: (1) MB-PDT at a fixed drug/light dose plus standard of care abscess drainage, (2) MB-PDT at a patient-specific dose determined by pre-treatment optical measurements plus standard of care abscess drainage, and (3) standard of care abscess drainage alone. The primary endpoint is time to removal of the drainage catheter. The secondary endpoint is reduction in bacterial burden from pre- to post-intervention. Tertiary endpoints include drain output following intervention, resolution of clinical symptoms, abscess recurrence, need for repeated intervention, and cure rate.

All subjects will receive standard of care image-guided percutaneous abscess drainage. This includes collection of a pre-intervention abscess aspirate sample, and placement of a drainage catheter.

For subjects in Arms 1 and 2, sterile methylene blue (MB) will then be administered to the abscess cavity using the same needle/catheter utilized for standard of care drainage. After a 10 minute incubation interval, MB will be aspirated and the cavity flushed with sterile saline.

For subjects in Arm 2, optical spectroscopy measurements will then be made to determine the optical properties of the abscess wall. This will be done by connecting the proximal end of the sterile optical fiber used for treatment illumination to a custom optical spectroscopy system. The distal end of this fiber will be advanced through the same catheter/needle used for the standard of care procedure in order to make gentle contact with the wall of the cavity. Low-intensity white light will be delivered by the fiber, and light that has interacted with the abscess wall will be detected by the same optical fiber. These optical measurements will be averaged and used to extract the absorption and reduced scattering coefficients at the treatment wavelength. These extracted optical properties, along with the subject's segmented pre-procedure CT images, will be used to generate a patient-specific treatment plan that seeks to deliver a desired fluence rate to 95% of the abscess wall, while limiting the portion of the abscess wall that receives a high fluence rate (>400 mW/cm2) to less than 5%.

For subjects in Groups 1 and 2, the cavity will then be filled with sterile 0.1% lipid emulsion solution to gently distend the cavity, and through efficient light scattering, homogenize the light dose to the walls of the cavity. A sterile optical fiber will be advanced to the approximate center of the abscess cavity via the same catheter/needle under image guidance. The proximal end of the fiber is coupled to the output of a diode laser system emitting light at 665 nm.

For subjects in Group 1 (MB-PDT at a fixed dose), laser power will be delivered to the cavity at a constant fluence rate. The laser power required to obtain the desired fluence rate at the wall will be calculated purely based on the abscess size. For subjects in Group 2 (MB-PDT with patient-specific treatment planning), the subject's measured optical properties and their segmented pre-procedure CT images will be integrated with treatment planning software to determine the laser power required to deliver the desired fluence rate to 95% of the abscess wall, while limiting the portion of the abscess wall that receives a fluence rate of >400 mW/cm2 to less than 5%. In both cases, illumination will be delivered for 20 minutes, resulting in a total delivered fluence of 24 J/cm2. Immediately after laser irradiation, the Intralipid solution will be aspirated and the cavity again flushed with sterile saline.

Collection of aspirated abscess material for microbiological assessment is standard of care for percutaneous abscess drainage. A portion of this standard of care collection will be collected by the study team for additional quantitative evaluation. Additionally, a post-intervention aspirate sample will be collected for study purposes.

If successful, this research could result in an adjunct treatment for abscess patients that improves long-term abscess resolution and the rate of response to percutaneous drainage. This clinical strategy would offer a wide range of potential health benefits to patients with deep tissue abscess. Among these advantages are reduced surgical intervention, decreased spread of infection, shortened course of post-treatment antibiotic therapy, and decreased selective pressure for antibiotic resistance. Ultimately, this would promote early recovery, shorten hospital stay, and lead to lower overall health care costs for patients undergoing image-guided percutaneous abscess drainage.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years or older
* All patients with clinical symptoms (ex: fever, chills, pain, tachycardia, hypotension), laboratory (leukocytosis) and radiologic findings (thick walled, rim-enhancing collection with gas bubbles or air-fluid levels) compatible with an abscess that requires image- guided percutaneous drainage
* Approval by the primary care team to pursue PDT and discuss enrollment with the patient

Exclusion Criteria:

* Pregnancy
* Lactation
* Allergy to contrast media, narcotics, sedatives, atropine or eggs
* Necrotic tissue that requires surgical debridement
* Severely compromised cardiopulmonary function or hemodynamic instability
* Thrombocytopenia (<50,000/mm3)
* Uncorrectable coagulopathy
* Poor kidney function (serum creatinine >3mg/dl)
* Lack of a safe pathway to the abscess or fluid collection
* Unable or unwilling to understand or to provide informed consent
* Unable or unwilling to undergo study procedures
* Patient unable to cooperate with, or to be positioned for the procedure
* Unable to comply with necessary follow up
* Patients with pancreatic abscesses
* Patients with known fistulous communication with their abscess
* Abscess greater than 13 cm in diameter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-07-15 (Estimated); Primary Completion 2031-06-30 (Estimated); Study Completion 2031-06-30 (Estimated)

PRIMARY OUTCOMES:
Time to removal of the drainage catheter | Day 1 post-intervention until removal of drainage catheter
  Drainage catheter output into the drainage bag will be noted daily by a member of the study team and the drainage catheter will be removed when output is reduced to <5 mL/day, as is standard of care for this patient population. Time to drainage catheter removal (in days) will be recorded for all subjects.

SECONDARY OUTCOMES:
Mean Change in bacterial burden | Pre and post intervention (approximately 24 hours)
  The outcome is reduction in colony-forming units per mL (CFU/mL) of bacteria in aspirate samples collected before and after intervention, measured on a log10 scale.
Total volume of catheter drainage output | day 14
  Daily output from the placed drainage catheter will be followed from the day of intervention to the either 14 days post-intervention or removal of the drainage catheter, whichever comes first. Daily drainage volume will be recorded, and cumulative drainage volume for the entire catheter placement will be reported.
mean number of days from intervention to symptom resolution | day 14
  Daily report of fever, chills, pain, heart rate, and blood pressure. The first day on which there is no report of fever, chill, or pain, and where heart rate and blood pressure are within normal ranges for the subject, will be recorded as the date of clinical symptom resolution. The mean number of days from intervention to symptom resolution will be recorded for each arm.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy M Baran, PhD, Principal Investigator — University of Rochester; Ashwani K Sharma, MD, Principal Investigator — University of Rochester; Laurie Christensen, BS, Study Director — University of Rochester
Locations (2):
- United States (2):
  - Highland Hospital, Rochester, New York
  - University of Rochester Medical Center, Rochester, New York

IPD SHARING:
Plan to Share IPD: No